CLINICAL TRIAL: NCT07057544
Title: The Role of Ultra-high-frequency ECG in the Localization of Left Ventricular Conduction Disorders and Prediction of Response to Resynchronization Therapy
Brief Title: UHF ECG in LBBB and Response to CRT Prediction
Acronym: UHF BLOCK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty Hospital Kralovske Vinohrady (Other Government)
Responsible Party: Principal Investigator, Karol Curila, MD, PhD, Faculty Hospital Kralovske Vinohrady
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UHFBLOCK trial; NW24-02-00143 (Other: Ministry of HealthCare of Czech Republic)
Record Dates: First submitted 2025-06-30; First posted 2025-07-10 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Left Bundle Branch Block; Left Bundle Branch Area Pacing; Biventricular Pacing; Intraventricular Conduction Delay
Keywords: left bundle branch block; resynchronization therapy; intraventricular conduction delay; left bundle branch pacing; biventricular pacing
MeSH Terms: conditions — Bundle-Branch Block

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CSP-CRT arm (Experimental): In this arm, LBBAP CRT will be performed
  Interventions: Device: LBBAP CRT device implantation
- BVP-CRT arm (Active Comparator): In this arm, BVP CRT will be performed.
  Interventions: Device: BVP-CRT

INTERVENTIONS:
Device: LBBAP CRT device implantation — Pacing system with a lead implanted in the left bundle branch area will be done.
  Arms: CSP-CRT arm
Device: BVP-CRT — Implantation of biventricular device
  Arms: BVP-CRT arm

SUMMARY:
The main objective of the project is to demonstrate that in patients with heart failure and QRS complex of nonRBBB morphology lasting over 130 ms, UHF-ECG can differentiate patients with trueLBBB from IVCD better than existing approaches based on the assessment of QRS complex morphology and duration from 12-lead ECG.

Another goal of the proposed study is to demonstrate that trueLBBB patients will benefit more from CRT using left bundle branch pacing than from CRT using biventricular pacing.

The final aim of the project is to demonstrate that the echocardiographic and clinical response in patients with intraventricular conduction disturbance will be dependent on the degree of reduction in ventricular dyssynchrony after CRT.

DETAILED DESCRIPTION:
Since the introduction of cardiac resynchronization therapy (CRT), a way to better define the patients who will benefit from it most has been sought. Their selection based on the duration of the QRS complex or its morphology fails in some of them. Current data demonstrate that CRT done by pacing the conduction system below the site of the left bundle branch block may be a better therapy than biventricular pacing. A prerequisite for a better effect of conduction system pacing is to perform it in patients in whom a conduction block is present in the left bundle branch block ("true" LBBB) and not in the patients with a more distal left ventricular conduction problem (IVCD). The criteria derived from the surface standard ECG are insufficient to differentiate "true" LBBB from IVCD, and thus it is not possible to determine the optimal treatment in some patients. The sequence of ventricular activation can be visualized within a few minutes using ultra-highfrequency ECG (UHF-ECG) in virtually all patients. It is a non-invasive method that shows ventricular dyssynchrony as a time difference between the activation of the ventricles or their individual segments. Pilot data show that patients with "true" LBBB are likely to have greater ventricular dyssynchrony and a different pattern of ventricular depolarization than patients with IVCD. The aim of this project is to test the hypothesis that UHF-ECG can distinguish "true" LBBB from IVCD in patients with heart failure and left ventricular conduction disturbance better than using standard criteria assessing QRS duration and morphology. Other aim is to demonstrate that in patients with trueLBBB resynchronization using conduction system pacing will lead to better echocardiographic and clinical outcomes than biventricular pacing. Finally, the echocardiographic and clinical response of IVCD patients will depend on the reduction of UHF-ECG ventricular dyssynchrony after CRT.

ELIGIBILITY:
Inclusion Criteria:

* HF due to ischemic or non-ischemic cardiomyopathy
* known coronary angiography
* NYHA II-IV
* LVEF ≤40%
* non-RBBB QRSd lasting >130 ms (by automated measurement)
* proximal LBBB proved by an invasive EP study or non-invasive dyssynchrony assessment in case such a method is confirmed to be non-inferior to an invasive EP study during the project

Exclusion Criteria:

* Age ˂18 years
* heart failure from reversible causes
* Moderate to severe aortic stenosis
* pregnancy
* active myocarditis
* hypertrophic cardiomyopathy
* cardiac valve surgery in the last three months
* myocardial infarction, PCI, or CABG in the last three months
* severe valvular disease requiring intervention
* severe atherosclerotic disease of the aorta and/or femoral arteries
* life expectancy ˂1 year
* known medical condition or contraindication causing potential complications for EP study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Left ventricular end-systolic volume | 6 and 18 months since randomization
  Left ventricular end-systolic volume reduction

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty Hospital Kralovske Vinohrady, Prague, Česká Republika, Czechia

IPD SHARING:
Plan to Share IPD: Undecided